CLINICAL TRIAL: NCT03645538
Title: Analysis of Cortical Biomarkers for Parkinson's Disease Patients
Brief Title: Analysis of Cortical Biomarkers for PD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Clinical professor, Universidade Federal de Pernambuco
Other Study IDs: Cortical_Biomarkers_EEG_ PD
Record Dates: First submitted 2018-07-25; First posted 2018-08-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease; Healthy
Keywords: Parkinson's disease; Healthy subjects
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Parkinson's disease patients: PD patients, after reading and signing the free and informed consent will be submitted to a single session to obtain the normal neurophysiological and behavioral endpoints and thus compare with those obtained in healthy individuals. All volunteers (healthy and patients) will be submitted to a behavioral and neurophysiological evaluation through transcranial magnetic stimulation (TMS) and electroencephalography (EEG).
  The neurophysiological evaluation will be conducted during "ON" (with medication) and "OFF" (without medication) period, by transcranial magnetic stimulation by single pulse (EMT-p) and by EEG.
  Interventions: Other: Parkinson's disease patients
- No drug - Control group: PD patients, after reading and signing the free and informed consent will be submitted to a single session to obtain the normal neurophysiological and behavioral endpoints and thus compare with those obtained in healthy individuals. All volunteers (healthy and patients) will be submitted to a behavioral and neurophysiological evaluation through transcranial magnetic stimulation (TMS) and electroencephalography (EEG).
  Interventions: Other: No drug

INTERVENTIONS:
Other: Parkinson's disease patients — The neurophysiological evaluation will be conducted during "ON" (with medication) and "OFF" (without medication) period, by transcranial magnetic stimulation by single pulse (EMT-p) and by EEG.
  Groups: Parkinson's disease patients
Other: No drug — The neurophysiological evaluation in healthy subjects will be conducted by transcranial magnetic stimulation by single pulse (EMT-p) and by EEG.
  Groups: No drug - Control group

SUMMARY:
Previous studies revealed changes in the pattern of cortical electrical activity of patients with Parkinson's disease (PD) and suggested that these changes may be dependent on the phenotypes of the disease and other related factors. A greater understanding of cortical electrical activity in PD patients may be relevant to guide professionals about the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). The present study aims to evaluate the pattern of brain activity of PD patients and to correlate the findings with the disease phenotypes and with other clinical characteristics. For this, volunteers with PD and healthy will participate in a single experimental session in which behavioral and electrophysiological assessments will be performed.

DETAILED DESCRIPTION:
Healthy individuals, after reading and signing the free and informed consent will be submitted to a single session to obtain the normal neurophysiological and behavioral endpoints and thus compare with those obtained in individuals with PD. All volunteers (healthy and patients) will be submitted to a behavioral and neurophysiological evaluation through transcranial magnetic stimulation (TMS) and electroencephalography (EEG).

The neurophysiological evaluation will be conducted during "ON" (with medication) and "OFF" (without medication) period, by transcranial magnetic stimulation by single pulse (EMT-p) and by EEG. TMS can perform different measures for the study of cortical excitability. The analysis of the motor cortex excitability will be held by: (i) determination of motor threshold (ii) the amplitude of the motor evoked potential (MEP). Since the assessment of the cortex activity will be held by: (i) power spectrum density (PSD) of all frequencies bands.75 For evaluation with the TMS (Neurosoft - Russia) volunteers will be instructed to sit in a chair and get comfortable position. Initially single TMS stimuli will be administered over the motor cortex to determine the cortical representation area of the first dorsal interosseous muscle (FDI) - MEP region whose response occurs more intensely observed by electromyography. The electrodes with 10 mm diameter should be placed on the belly of the target muscle and the reference electrode is placed in the interphalangeal joint of the thumb. All care for the acquisition of electromyographic signal will be taken according to the criteria of Surface Electromyography for the Non-invasive Assessment of Muscles (SENIAM).

For the location of the representative FDI muscle cortical region coil with an angle of 45 degrees is positioned at a distance of 20% of Cz point (according to the international system for marking 10-20) bring into the contralateral muscle to be evaluated. For all evaluations the same coil is used, the figure-eight angled in order to avoid measurement bias. To assess cortical excitability of both hemispheres, the following measures are carried out: resting motor threshold (RMT) and motor evoked potentials (MEP).

For EEG assessment, the electrodes will be positioned on the scalp of the individual, according to the international 10-20 marking system, maintained with the maximum impedance of 10kΩ. During the acquisition of the electroencephalographic signal, a motor imagery and execution protocol will be performed, in both upper limbs. The collected data will be further processed and analyzed by MATLAB® software for Windows.

For behavioral assessment the following scales and tests will be performed during "ON" (with medication) and "OFF" (without medication) period: Parkinson's disease sleep scale; Geriatric Depression Scale; Edinburgh Handedness Inventory; International Physical Activity Questionnaire; Timed up and go test; Berg Balance Scale; Unified Parkinson's disease Rating Scale sessions II and III.

ELIGIBILITY:
Inclusion Criteria:

* · Ages: 40 years or greater

  * Gender: Both
  * Minimum score of the Montreal Cognitive Assessment (MoCA) (27 points);
  * Regular antiparkinsonian pharmacological treatment;
  * Staged from I to IV on the modified Hoehn & Yahr scale.

Healthy Subjects inclusion criteria:

* Ages: 40 years or greater
* Gender: Both
* Subjects who do not have self-report of neurological or articular disorder

Exclusion Criteria:

* · Pregnant women;

  * Pacemaker;
  * History of seizures;
  * Metallic implants in the head;
  * Patients with clinical evidence of brain injuries;
  * Individuals with other neurological disorders, postural hypotension, vestibular, visual, cardiovascular or musculoskeletal disorders that affect the performance of the proposed tests;
  * Other diseases in lower limbs that interfere with performance and locomotion;
  * Submitted to previous surgical intervention for PD.

Healthy Subjects exclusion criteria:

* Pregnant women;
* Pacemaker;
* History of seizures;
* Metallic implants in the head;
* Patients with clinical evidence of brain injuries;
* Chronic pain associated to other diseases;
* Use of neuroleptic medications
* Individuals with other neurological disorders, postural hypotension, vestibular, visual, cardiovascular or musculoskeletal disorders that affect the performance of the proposed tests.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be invited to participate in the study from broad divulgation of research through print and digital media. Volunteers with PD and healthy who meet the inclusion and exclusion criteria of the study will be selected by means of non-probabilistic sampling.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in cortical activity | before and 1 hour after the medication ingestion.
  For EEG assessment, the electrodes will be positioned on the scalp of the individual, according to the international 10-20 marking system, maintained with the maximum impedance of 10kΩ. During the acquisition of the electroencephalographic signal, a motor imagery and execution protocol will be performed, in both upper limbs. The collected data will be further processed and analyzed by MATLAB® software for Windows.

SECONDARY OUTCOMES:
Change in motor threshold | before and 1 hour after the medication ingestion.
  to determine the resting motor threshold (RMT), the minimum of stimulator output necessary to emit 5 pulses with amplitudes above 50 microvolts in 10 trials. The investigators will use the motor threshold assessment tool to perform RMT assessment. Motor threshold means a measure of pyramidal neurons.
Change in motor evoked potentials | before and 1 hour after the medication ingestion.
  to measure the MEP, the intensity of the magnetic stimulator will be adjusted to 120% of RMT and 20 stimuli will be registered. The volunteer will be sitted, completely relaxed. The amplitude means of evoked potentials will determine the MEP.

OTHER OUTCOMES:
Change in functional mobility | before and 1 hour after the medication ingestion.
  The evaluation of the basic functional mobility of individuals will be performed by the Timed up and go test. It is analyzed the time spent by the individual to get up from a chair with arms, walk for three meters and return to the chair. Higher time values and step numbers represent a greater risk of falls.
Change in balance | before and 1 hour after the medication ingestion.
  The balance of individuals will be assessed through the Berg Balance Scale, which comprises 14 items with a score of 0-4 each from 0 (worst) to 4 (best performance), used to assess dysfunction in balance and independence in life activities daily.
Change in motor impairment | before and 1 hour after the medication ingestion.
  The Unified Parkinson's disease rating scale (UPDRS) will be applied to assess the motor performance of individuals. It is the most commonly used scale for assessing the severity of PD. In the present study, the UPDRS session III will be analyzed, comprising 14 items with a score of 0-4 each, from the best to the worst motor performance. According to the scores presented in UPDRS, patients will be classified as: (i) tremor-dominant or (ii) with postural instability and gait difficulty.
Sleep quality | before the medication ingestion.
  PDSS is composed by 15 questions that assess nocturnal disorders caused by PD symptoms, whose scores vary from 0 (zero), considered as the worst perception of sleep quality, and 10 (ten) the best. Overall scores less than 82 or less than five in each subitem may be indicative of changes in sleep quality
Depression level | before the medication ingestion.
  The scale is one of the most sensitive and reliable for the detection of depression in the elderly and PD patients. It is a 30-question scale that assesses the individual's perception of their feelings in the last week. Individuals can be classified according to the following extracts: absence of depression (0-9 points); mild depression (11-20 points); severe depression (21-30 points).
Handedness | before the medication ingestion.
  For the determination of the handedness, the Edinburgh Handedness Inventory will be used, consisting of 10 questions about the manual preference in performing 10 tasks usually performed by most people. Positive values are considered for the right hand and negative for the left hand. A score of +10 points will be awarded if the patient performs activity exclusively with the right hand and -10 points if performed exclusively with the left. For activities performed with both hands, +5 points to the right and -5 points to the left, the inventory can total 100 positive or negative points. The sum is represented by the manual preference index, which should be> 70 if right dominance and ≤ -70 if left dominance.
Physical activity level | before the medication ingestion.
  To assess the level of physical activity performed by the individual, including daily and occupational tasks, the International Physical Activity Questionnaire (IPAQ) will be applied. The long version has 27 questions, subdivided into four dimensions of physical activity (work, transportation, domestic activities and leisure) and a session related to the time released sitting during the week. Individuals who perform physical activity within the current recommendation (at least 30 minutes a day, most days of the week), with the sum of at least 150 minutes per week of at least moderate intensity physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Lívia Shirahige, MsC, Principal Investigator — Universidade Federal de Pernambuco; Adriana Maciel, MsC, Study Chair — Universidade Federal de Pernambuco; Déborah Oliveira, MsC, Study Chair — Universidade Federal de Pernambuco; Fernanda Nogueira, Bachelor, Study Chair — Universidade Federal de Pernambuco; Marina Berenguer, Bachelor, Study Chair — Universidade Federal de Pernambuco; Brenda Valença, Study Chair — Universidade Federal de Pernambuco; Rodrigo Brito, Bachelor, Study Chair — Universidade Federal de Pernambuco
Locations (1):
- Applied Neuroscience Laboratory, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No